CLINICAL TRIAL: NCT02886910
Title: Chorioamnionitis: Observation of at Risk Infants vs Standard Care. Randomized Controlled Trial.
Brief Title: Chorioamnionitis: Observation of at Risk Infants vs Standard Care
Acronym: CHORIS-RCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Luca Ronfani, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC 18/14
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Chorioamnionitis; Early Onset Neonatal Sepsis; Sepsis of the Newborn
Keywords: Chorioamnionitis; Early onset neonatal sepsis; Antibiotics; Clinical observation
MeSH Terms: conditions — Chorioamnionitis; Neonatal Sepsis | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical observation (Experimental): Asymptomatic newborns born at term to mothers with suspected chorioamnionitis. They will receive a limited evaluation (blood culture, complete blood count), and a clinical observation. Antibiotics will be started only if sepsis-related signs or symptoms are present.
  Interventions: Other: Clinical observation
- Standard management (Active Comparator): Asymptomatic newborns born at term to mothers with suspected chorioamnionitis. The will receive a limited evaluation (blood culture, complete blood count), a clinical observation and antibiotics at birth.
  Interventions: Other: Clinical observation; Other: Standard management

INTERVENTIONS:
Other: Clinical observation — Antibiotics will be started only if sepsis-related signs or symptoms are present.Clinical observation consists in a standardized physical examination protocol according to which newborns are observed by the nurses at 1, 2, 4, 8, 12, 16, 20, 24 hours of life and then every 6 hours up to 48 hours of life. The following signs and symptoms are checked: skin colour (pink/pale/cyanotic/mottled), respiratory rate (lower or higher than 60 breaths/minute) and presence or absence of respiratory distress.
Other: Standard management — Antibiotics will be started at birth. Clinical observation will be carried out with the same timing and protocol
  Arms: Standard management

SUMMARY:
This study evaluates the non-inferiority of a protocol of limited evaluation (complete blood count, blood culture) and clinical observation by standardized physical examination versus the algorithm suggested in the CDC's 2010 guidelines (limited evaluation, clinical observation and antibiotic therapy) in the management of asymptomatic infants born at term to mothers with suspected chorioamnionitis. The primary outcome of the study is the difference in the prevalence of sepsis-related symptoms between the two groups.

DETAILED DESCRIPTION:
Chorioamnionitis complicates 1-3% of pregnancies at term. The current international guidelines of the Center for Disease Control (CDC 2010) recommend that all asymptomatic newborns born to mothers with suspected chorioamnionitis undergo limited evaluation (i.e. blood culture at birth and complete blood count) and antibiotic therapy until the blood culture result is available.

However, the prevalence of positive blood cultures in infants born to mothers with suspected chorioamnionitis is low, approximately 1%, including also infants requiring intensive care. This prevalence is even lower in asymptomatic infants. Moreover, the efficacy of antibiotic prophylaxis in preventing early sepsis, death or long-term sequelae in asymptomatic infants born to mothers with suspected chorioamnionitis has not been demonstrated.

Early antibiotic use has been related to obesity and to the modification of microbiota. Limiting antibiotic use may prevent the emergence of antibiotic-resistant bacteria.

Clinical observation is a reliable method to recognize infants with sepsis.

ELIGIBILITY:
Inclusion Criteria:

- asymptomatic newborns born at term (>= 37 weeks of gestational age)

Exclusion Criteria:

* preterm newborns (< 37 weeks gestational age)
* sepsis-related signs of symptoms at birth
* intensive care admittance

Ages: 10 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Sepsis-related signs and symptoms | 48 hours of life
  Presence of pale/cyanotic/mottled skin, respiratory rate higher than 60 breaths/minute or respiratory distress

SECONDARY OUTCOMES:
Mortality | 21 days
Neonatal intensive care unit admittance | 21 days
Days of antibiotics | 21 days
Days of hospitalization | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Demarini, MD, Study Director — Institute for maternal and child health - IRCCS "Burlo Garofolo", Trieste, Italy
Locations (1):
- Institute for Maternal and Child Health IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No